CLINICAL TRIAL: NCT03435796
Title: Long-Term Follow-up Protocol for Subjects Treated With Gene-Modified T Cells
Brief Title: Long-Term Follow-up Protocol for Participants Treated With Gene-Modified T Cells
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GC-LTFU-001; U1111-1206-8250 (Registry Identifier: WHO); 2023-504201-36 (Other: EU CTR)
Record Dates: First submitted 2018-01-09; First posted 2018-02-19 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Neoplasms
Keywords: Long-term follow up; Gene-Modified T Cells; CAR T Cell
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants exposed to Gene-modified (GM) T cell therapy (Other)
  Interventions: Genetic: Gene-modified (GM) T cell therapy

INTERVENTIONS:
Genetic: Gene-modified (GM) T cell therapy — No investigational product will be administered

SUMMARY:
This is a prospective study for the long-term follow-up (LTFU) of safety and efficacy for all pediatric and adult participants exposed to Gene-modified (GM) T-cell therapy participating in a previous Celgene sponsored or Celgene alliance partner sponsored study.

Participants who received at least one infusion of GM T cells will be asked to enroll in this LTFU protocol upon either premature discontinuation from, or completion of the prior parent treatment protocol.

ELIGIBILITY:
Inclusion Criteria:

* Received at least one gene-modified (GM) T-cell infusion in a previous Celgene sponsored, Juno Therapeutics, other affiliates of BMS, or Celgene alliance partner-sponsored trial, and have discontinued, or completed the post-treatment follow-up period in the parent treatment protocol, as applicable.
* Must understand and voluntarily sign an Informed Consent Form/Informed Assent Form prior to any study-related assessments/procedures being conducted.

Exclusion Criteria:

Not Applicable

Other protocol-defined inclusion/exclusion criteria apply

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1541 (Estimated)
Dates: Start 2018-07-19 (Actual); Primary Completion 2036-11-30 (Estimated); Study Completion 2036-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of delayed Adverse Events (AEs) | Up to 15 years from last gene-modified (GM) T cell infusion
Persistence of GM T cell drug products | Up to 15 years from last GM T cell infusion
Analysis of vector integration sites | Up to 15 years from last GM T cell infusion
Incidence of replication-competent lentiviruses | Up to 15 years from last GM T cell infusion
Physical growth as assessed by physical examination (pediatric participants only) | Up to 15 years from last GM T cells infusion or until Tanner Stage 5 is reached
Incidence of sexual maturation as assessed by the Tanner staging system (pediatric participants only) | Up to 15 years from last GM T cells infusion or until Tanner Stage 5
Proportion of participants who progressed on the study: participants with original diagnosis of malignancies | Up to 15 years from last GM T cells infusion
Overall Survival (participants with original diagnosis of malignancies) | Up to 15 years from last GM T cells infusion

SECONDARY OUTCOMES:
Lymphocyte count (B-cell) | Up to 15 years
  If B-cell recovery criteria are not met at Month 60 (Year 5), then annual monitoring will continue up to 15 years, until subject withdrawal of consent, or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (191):
- United States (97):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic Phoenix, Phoenix, Arizona
  - Arizona Cancer Center, Scottsdale, Arizona
  - Local Institution - 01021, Tucson, Arizona
  - City Of Hope, Duarte, California
  - University Of California San Diego Moores Cancer Center, La Jolla, California
  - Local Institution - 01206, Los Angeles, California
  - Local Institution - 01043, Sacramento, California
  - University of California, San Francisco- California, San Francisco, California
  - UCLA Medical Centre-Santa Monica, Santa Monica, California
  - Stanford Cancer Center, Stanford, California
  - University Of Colorado Cancer Center, Aurora, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Local Institution - 01050, Washington D.C., District of Columbia
  - The Mayo Clinic - Jacksonville, Davis-E, Jacksonville, Florida
  - Baptist Cancer Center, Miami, Florida
  - Local Institution - 01035, Orlando, Florida
  - H. Lee Moffitt Cancer Center and Research Institute University of South Florida, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Northside Hospital, Inc, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University Of Chicago Medical Center, Chicago, Illinois
  - Local Institution - 01040, Maywood, Illinois
  - Local Institution - 01063, Niles, Illinois
  - IN Univ Simon Cancer Center, Indianapolis, Indiana
  - Local Institution - 01020, Indianapolis, Indiana
  - Kansas University Medical Center, Westwood, Kansas
  - Cancer Center of Kansas, Wichita, Kansas
  - University Of Kentucky, Lexington, Kentucky
  - Norton Cancer Institute Louisville Oncology, Louisville, Kentucky
  - Local Institution - 01026, New Orleans, Louisiana
  - University of Maryland - Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Sidney Kimmel Comp Cancer Center at Johns Hopkins, Baltimore, Maryland
  - National Cancer Institute, Bethesda, Maryland
  - Local Institution - 01107, Boston, Massachusetts
  - Massachusetts General Hospital / Dana-Farber Cancer Institute, Boston, Massachusetts
  - Local Institution - 01106, Boston, Massachusetts
  - University Of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Karmanos Cancer Center Wayne State University, Detroit, Michigan
  - Providence Cancer Institute, Southfield, Michigan
  - M Health Fairview University of Minnesota Medical Center - East Bank, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Siteman Cancer Center, St Louis, Missouri
  - University Of Nebraska Medical Center, Omaha, Nebraska
  - Local Institution - 01030, East Brunswick, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Memorial Hosp, Morristown, New Jersey
  - Local Institution - 01053, New Brunswick, New Jersey
  - New York Oncology Hematology P.C., Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Local Institution - 01066, New York, New York
  - Weill Cornell Medicine / New York Presbyterian Hospital, New York, New York
  - Icahn School Of Medicine At Mount Sinai, New York, New York
  - Columbia University Medical Center/New York-Presbyterian Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Local Institution - 01051, Rochester, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Novant Health, Salisbury, North Carolina
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center (OSUCCC) - The James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - University of Oklahoma Peggy and Charles Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Willamette Valley Cancer Institute, Eugene, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Oregon Health and Science University OHSU, Portland, Oregon
  - Children's Hospital of Philadelphia-Center for Childhood Cancer Research, Philadelphia, Pennsylvania
  - University of Pennsylvania Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Thomas Jefferson University - Clinical Research Institute, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC Cancer Pavillion, Pittsburgh, Pennsylvania
  - Hematology and Oncology Associates of SC, LLC, Greenville, South Carolina
  - Local Institution - 01064, Sioux Falls, South Dakota
  - Sarah Cannon Research Inst, Nashville, Tennessee
  - Texas Oncology, Dallas, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - University of Texas- MD Anderson, Houston, Texas
  - Sam Clinical Research Center, San Antonio, Texas
  - Local Institution - 01033, Temple, Texas
  - Texas Oncology, P.A. - Tyler, Tyler, Texas
  - University of Utah - Huntsman Cancer Institute, Salt Lake City, Utah
  - Intermountain Healthcare - LDS Hospital, Salt Lake City, Utah
  - University Of Virginia Health System, Charlottesville, Virginia
  - Local Institution - 01045, Norfolk, Virginia
  - Local Institution - 01023, Richmond, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - Local Institution - 01060, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Local Institution - 01055, Tacoma, Washington
  - University Of Wisconsin, Madison, Wisconsin
  - Froedtert Hospital BMT Medical College of Wisconsin, Milwaukee, Wisconsin
  - Local Institution - 01069, Wauwatosa, Wisconsin
- Australia (3):
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Allgemeinen Krankenhaus (AKH) Wien - Medizinische Universitaet Wien, Vienna, Austria
- Belgium (6):
  - Jules Bordet Institut, Anderlecht
  - Universitair Ziekenhuis Brussel, Brussels
  - Local Institution - 05200, Ghent
  - Uz Gent, Ghent
  - University Hospital Leuven, Leuven
  - Local Institution - UNK 2, Leuven
- Canada (5):
  - University Of Calgary, Calgary, Alberta
  - Local Institution - 02802, Vancouver, British Columbia
  - Local Institution - 02801, Hamilton, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - CIUSSS de l'Est-de-l'Ile-de-Montreal, Montreal, Quebec
- Helsinki University Central Hospital (HUCH), Helsinki, Finland
- France (15):
  - Hopital Henri Mondor, Creteil-Paris
  - CHRU de Lille France, Lille
  - Local Institution - 09601, Lyon
  - Local Institution - 09400, Marseille
  - Local Institution - 09602, Marseille
  - CHU Montpellier - Hôpital Saint Eloi, Montpellier
  - Chu Hotel Dieu, Nantes
  - Hopital Saint Louis, Paris
  - Hospital Saint Louis, Paris
  - Local Institution - 09600, Paris
  - Centre Hospitalier Universitaire (CHU) de Bordeaux - Hopital Haut-Leveque, Pessac
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - CHU La Miletrie, Poitiers
  - Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse
  - Gustave Roussy, Villejuif
- Germany (13):
  - Robert-Rossle-Klinik im HELIOS Klinikum Berlin-Buch Klinik fur Hamatologie, Onkologie u. Tumorimmuno, Berlin
  - Local Institution - 03155, Berlin
  - Kinikum der Universitaeat zu Koeln, Cologne
  - Universitatsklinikum Carl Gustav Carus an der TU Dresden, Dresden
  - Local Institution - 03513, Düsseldorf
  - Local Institution - 03500, Frankfurt
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Universitatsklinikum Heidelberg, Heidelberg
  - LMU Klinikum der Universität, München
  - Local Institution - 03454, Münster
  - Local Institution - 03503, Tübingen
  - University Hospital of Ulm, Ulm
  - Universitatsklinikum Wurzburg Medizinische Klinik und Poliklinik II, Würzburg
- Israel (2):
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
  - The Chaim Sheba Medical Center, Tel Litwinsky
- Italy (10):
  - Ospedali Riuniti di Ancona, Ancona
  - Azienda Ospedaliero Universitaria Di Bologna Policlinico Sorsola Malpighi, Bologna
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Fondazione Monza e Brianza per il Bambino e la sua Mamma (MBBM), Monza
  - Istituto Nazionale Per Lo Studio E La Cura Dei Tumori Fondazione Giovanni Pascale, Naples
  - Local Institution - 07500, Roma
  - Ospedale Pediatrico Bambino Gesu, Rome
  - Istituto Clinico Humanitas, Rozzano (MI)
  - Local Institution - 07610, Torino
  - Azienda Sanitaria Ospedaliera San Giovanni Battista Molinette, Turin
- Japan (11):
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Toranomon Hospital, Minato-ku, Tokyo
  - Local Institution - 13202, Bunkyō City
  - Kyushu University Hospital, Fukuoka
  - Tokai University Hospital, Isehara City, Kanagawa
  - Nagoya City University Hospital, Nagoya
  - Osaka Metropolitan university Hospital, Osaka
  - Japan Red Cross Medical Center, Shibuya-ku
  - Local Institution - 13804, Shinjuku
- Netherlands (3):
  - Local Institution - 04650, Amsterdam
  - Erasmus Medical Center - Daniel den Hoed, Rotterdam
  - Local Institution - 04400, Utrecht
- Oslo Universitetssykehus, Oslo, Norway
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - St Johns Cancer Centre in Lublin, Lublin
  - Instytut Hematologii I Transfuzjologii, Warsaw
- Institutul Clinic Fundeni, Bucharest, Romania
- South Korea (3):
  - Asan Medical Center (AMC), Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (9):
  - Hospital Universitario Vall D hebron, Barcelona
  - Hospital Universitari Germans Trias i Pujol ICO Badalona, Barcelona
  - Institut Clinic de Nefrologia i Urologia - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital San Joan de Deu Barcelona, Esplugues de Llobregat
  - Hospital Infantil Universitario Nino Jesus, Madrid
  - Hospital 12 De Octubre, Madrid
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Universitario de Salamanca - Complejo Asistencial Universitario de Salamanca, Salamanca
  - Hospital Virgen Del Rocio, Seville
- Karolinska University Hospital Huddinge, Stockholm, Sweden
- Inselspital Bern, Bern, Switzerland
- United Kingdom (5):
  - Local Institution - 10850, Leeds
  - Kings College Hospital, London
  - UCL Cancer Institute, London
  - Christie Hospital Nhs Trust, Manchester Withington
  - Somers Cancer Research Building, Shirley Southampton

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- [Derived] Abramson JS, Palomba ML, Gordon LI, Lunning M, Wang M, Arnason J, Purev E, Maloney DG, Andreadis C, Sehgal A, Solomon SR, Ghosh N, Dehner C, Kim Y, Ogasawara K, Kostic A, Siddiqi T. Two-year follow-up of lisocabtagene maraleucel in relapsed or refractory large B-cell lymphoma in TRANSCEND NHL 001. Blood. 2024 Feb 1;143(5):404-416. doi: 10.1182/blood.2023020854. PMID 37890149
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html